CLINICAL TRIAL: NCT01301404
Title: Oral Rehydration Therapy With 10% Carbohydrate Drink for Preventing Postoperative Nausea and Vomiting (PONV) After Low Dose of Spinal Morphine in Patients Undergoing Total Knee Replacement
Brief Title: 10% Carbohydrate Drink for Preventing Post-operative Nausea and Vomiting (PONV) After Spinal Morphine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Manee Raksakietisak, Associate professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 763/2553(EC2)
Record Dates: First submitted 2011-02-20; First posted 2011-02-23 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2012-06

CONDITIONS: Nausea and Vomiting, Postoperative
Keywords: Postoperative nausea and vomiting (PONV); Spinal morphine; Total knee replacement (TKR); blood sugar; carbohydrate drink
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): patient receive nothing
- carbohydrate drink (Experimental): 10%carbohydrate drink
  Interventions: Dietary Supplement: 10% carbohydrate drink

INTERVENTIONS:
Dietary Supplement: 10% carbohydrate drink — In the study group, 10% carbohydrate drink 400 ml will be given between 18-24 hr the night before surgery and another 400 ml will be drunk at 6-7 hr in the morning of surgery.
  Other Names: Green mate (orange favor)
  Arms: carbohydrate drink

SUMMARY:
PONV after intrathecal morphine, occurs up to 30-40 percent. The patients having TKR normally are female, obese and non-smoker which are risk factors for PONV. Recently, a multimodal approach, combining several means to minimize PONV, has found wide acceptance as a standard of care. In our hospital, most of the patients are supposed to fast after midnight The oral rehydration therapy reduce patients thirst and increase his satisfaction, but whether or not this method can reduce the incidence of PONV after low dose (0.2 mg) intrathecal morphine is not investigated yet. The aim of this study is to investigate the effect of preoperative oral rehydration therapy on the incidence of PONV.

DETAILED DESCRIPTION:
We enroll patients who are undergoing TKR under spinal anesthesia with 0.5% heavy bupivacaine 10-15 mg (2.0-3.0 ml)+ intrathecal morphine 0.2 mg+ femoral nerve block with 0.25% bupivacaine 20 ml.

The enrolled patients will fast after midnight and in the morning they are allowed to drink 10% carbohydrate drink or not to drink (according to their randomization). 400 ml of 10% carbohydrate drink is drunk between evening and midnight and extra water if needed in the study group. In the control group, the patients are allowed to drink until midnight. Total of water consumption between 18.00-24.00 will be recorded in both groups. In the morning, the study group will drink another 400 ml of 10% carbohydrate drink between 6 - 7 am. The premedications should not include sedation or GI mobility drugs. Before starting anesthesia, the patients will be asked some questions about thirsty, hungry, anxiety and nausea and weigh their feeling from 0-10.

The surgery and pain therapy will be tha same in both groups and the PONV (incidence, severity and rescue therapy) at recovery room and 24 hours postoperative period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients are under going unilateral TKR, with ASA I-III who scheduled started in the morning list (before noon)

Exclusion Criteria:

* Diabetes
* History of motion sickness
* Chronic kidney disease (CKD, creatinine > 2 mg/dl)
* Hiatus hernia or gastro esophageal reflux
* Patients receiving drugs that might affect GI motility such as opioids

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative nausea and vomiting after TKR | 24 hours
  Compare the incidence, severity and rescue therapy of PONV in control (fast)group a group and the study (carbohydrate drink) group

SECONDARY OUTCOMES:
Incidence of hyperglycemia during perioperative period | 24 hours
  Regarding to the perioperative stress and carbohydrate drinking, we also measure blood sugar before and postoperation and compare their values between groups

CONTACTS AND LOCATIONS:
Overall Officials: Manee Raksakietisak, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand